CLINICAL TRIAL: NCT04853615
Title: Is SGLT2 Inhibitors a Better Prophylactic Agent Against Post-contrast Acute Kidney Injury in Diabetic Kidney Disease? A Multicenter Prospective Randomized Controlled Study
Brief Title: SGLT2 Inhibitors Prophylaxis Against Post-contrast Acute Kidney Injury in Diabetic Kidney Disease?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fayoum University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelkawi Hammad, Lecturer of internal medicine, Fayoum University
Other Study IDs: EC 2119
Record Dates: First submitted 2021-04-17; First posted 2021-04-21 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: SGLT2i Kideny Protection Against Contrast in Diabetic Kidney
MeSH Terms: interventions — empagliflozin; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: 1st group will receive normal saline 10ml/kg over 6 hours before and 6 hours after radiocontrast
- Group 2: 2nd group will receive allopurinol 300 mg and linagliptin 5 mg once daily
- Group 3: 3rd group will receive the SGLT2i empagliflosin 25 mg once daily
  Interventions: Drug: Empagliflozin 25 MG
- Group 4: 4thwill receive allopurinol and empagliflosin.
  Interventions: Drug: Empagliflozin 25 MG

INTERVENTIONS:
Drug: Empagliflozin 25 MG — PAtient will receive empagliflozin 25 mg daily
  Other Names: SGLT2 inhibitors
  Groups: Group 3; Group 4

SUMMARY:
We will look for the possible effect of SGLT2i as a single agent to prevent post-contrast Acute Kidney Injury in diabetic kidney disease.

DETAILED DESCRIPTION:
Population of Study o Group 1 :

1. st group will receive normal saline 10ml/kg over 6 hours before and 6 hours after radiocontrast.

   o Group 2 :
2. nd group will receive allopurinol 300 mg and linagliptin 5 mg once daily

   o Group 3 :
3. rd group will receive the SGLT2i empagliflosin 25 mg once daily

   o Group 4 :
4. thwill receive allopurinol and empagliflosin.

Inclusion Criteria :

o Age: more than30years, diabetes,diabetic kidney disease,GFR: more than30ml/min/1.73m2

Exclusion Criteria :

o Diabetics Patients with GFR less than 30 mL/min/1.73 m2.

Sample Size ( number of participants included ) :

800 patients Fayoum University Faculty of Medicine Scientific Research Ethics Committee

Methodology in details :

The chosen patients will be randomly allocated to 4 equal groups that will receive their prophylaxis for 48 hours before and 48 hours after the radiocontrast administration. Baseline serum creatinine will be obtained 72 hours before the planned intervention and before administration of any protective protocol and follow-up serum creatinine will be obtained 72 hours and 1 week after contrast administration. The first control group will receive normal saline 10ml/kg over 6 hours before and 6 hours after radiocontrast. Saline should be given by infusion pump to guarantee steady rate of infusion. 2nd group will receive allopurinol 300 mg and linagliptin 5 mg once daily. 3rd group will receive the SGLT2i empagliflosin 25 mg once daily, and the 4th will receive allopurinol and empagliflosin.

ELIGIBILITY:
Inclusion Criteria:

* Age: more than30years, Diabetes, Diabetic kidney disease, GFR: more than30ml/min/1.73m2

Exclusion Criteria:

* Diabetics Patients with GFR less than 30 mL/min/1.73 m2.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The chosen patients will be randomly allocated to 4 equal groups that will receive their prophylaxis for 48 hours before and 48 hours after the radiocontrast administration
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
SGLT2i proves protective effect | 72hours after contrast
  SGLT2i shows protected the kidneys against contrast injury

SECONDARY OUTCOMES:
SGLT2i is non inferior to allopurinol | 72hours after contrast
  SGLT2i showed noninferiorty whencompared to allopurinol

IPD SHARING:
Plan to Share IPD: Undecided